CLINICAL TRIAL: NCT05159856
Title: Early Detection of Long-term Diabetic Complications in Children and Adolescents With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Steno Diabetes Center Sjaelland (Other Government)
Responsible Party: Sponsor
Other Study IDs: H-20038547
Record Dates: First submitted 2021-11-15; First posted 2021-12-16 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Complications; type1diabetes; Children, Only; Diabetic Neuropathies; Arterial Stiffness
Keywords: pediatric; arteriel stiffness; pulse wave velosity; neuropathy; type 1 diabetes; early diabetic complications
MeSH Terms: conditions — Diabetes Complications; Diabetic Neuropathies; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — routine tests (hemoglobin and iron metabolites, BS, HbA1c, electrolytes, creatinine, urea, LDL, HDL, triglycerid, total cholesterol), and markers of glucose- (insulin, c-peptide), lipid- (leptin, adiponectin) bone- (VitD, calcium, PTH, phosphate, magnesium, BASP, OCN, P1NP, CTX, uOCN, sclerostine, RANKL., Osteoprotegrin and osteoglycin), gastrointestinal (GLP-1, GIP and glucagon). IGF-1 IGF-BP3, thyroid metabolism (TSH, T3, free T4), sex hormones, adrenal androgens, aldosterone and metabolomics.
  DNa for snp (single nucleotide polymorphisms) and HLA analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective cohort study (observational): 400 children/adolescents, aged 6-18 years, with type 1 diabetes for more than 12 months

SUMMARY:
Aims: To investigate early markers of long-term diabetic complications and the association to an extended glucose metabolic profile comprising glucose control (current and past), glucose variability and insulin sensitivity in children and adolescents with type 1 diabetes (T1D).

Background: Most Danish children and adolescents with T1D do not achieve their metabolic target and are at increased risk of developing long-term diabetic complications, reducing their life expectancy and increase their morbidity rate. Hence, improved metabolic control, a better understanding of what optimal metabolic control means, combined with detailed monitoring of the first markers of long-term complications and their reversibility or lack thereof are needed.

Methods: A prospectivel study of 400 children, aged 6-18 years old, with T1D>12 months. Early markers of long-term diabetic complications will be investigated as arterial stiffness, nerve dysfunction and nephropathy. Data on T1D onset, duration, treatment modality, self-monitoring-blood-glucose profiles, growth, weight, and pubertal status will be collected.

Blood sampling will include routine tests and markers of glucose, lipid, bone, and gastrointestinal metabolism. DXA-scan, Fibroscan, bone-age, eye-examination and physical activity will be measured. Data on retrospective glucose- and lipid-profiles will be collected. The children will be offered a followup every 5 years for the next two decades.

Perspectives: This study provides novel insight into the frequency of early markers of long-term diabetic complications and its association to the interplay of the pancreas, adipose, gastrointestinal and bone metabolic axis. Which can assist in identifying subgroups of children and adolescents requiring earlier in-depth screening for early markers of long-term diabetic complications, for putative interventions for prevention, hence reducing morbidity and mortality in T1D.

DETAILED DESCRIPTION:
The project is designed as a cross-sectional cohort study. The study consists of a one-day visit where 400 children and adolescents with T1D will be thoroughly examined after an overnight fast.

The following examinations are parof this study:

- Standard physical examination: Including cor/pulm/abdomen, heart rate and blood pressure measurement. Data regarding age, sex, diabetes duration, growth, weight, and pubertal status.

Blood sampling

* Bloodsampling: Include routine tests (hemoglobin and iron metabolites, BS, HbA1c, electrolytes, creatinine, urea, LDL, HDL, triglyceride, total cholesterol), and markers of glucose (insulin, c-peptide), lipid (leptin, adiponectin), bone (VitD, calcium, PTH, phosphate, magnesium, BASP, OCN, P1NP, CTX, uOCN, sclerostine, RANKL, osteoprotegrin and osteoglycin), gastrointestinal (GLP-1, GIP and glucagon) metabolism. IGF-1, IGF-BP3, thyroid metabolism (TSH, T3, free T4), sex hormones, adrenal androgens, aldosterone. Thyroid and celiac disease autoantibodies. Markers for inflammation and endothelial dysfunction will be examined. Plasma, serum and urine will also be collected for a Biobank for future research e.g. for studying metabolomics.
* Carotid-femoral pulse wave velocity: Assessed with the Sphygmocor (AtCor Medical) device to measure arterial stiffness in the large arteries.
* Evaluation of the nervous system function:
* Cardiac autonomic neuropathy function will be assessed by the Vagus device.
* Large sensory nerve function test assessed by sural nerve conduction velocity and sural nerve amplitude, measured with the non-invasive handheld device DPNCheckTM (NeuroMetrix, Inc., Waltham, USA).
* Small sympathetic nerve fiber function assessed by electrochemical skin conductance assessed using the non- invasive device Sudoscan™ (Impeto Medical, Paris, France).
* Kidney: Three morning urine samples will be collected at home for analyses of albumin/creatinine ratio.
* Bone age Measured on an x-ray of the left hand using BoneXpert software to adjust for potentially biological age.
* Dual energy X-ray absorptiometry scan: Performed to evaluate body composition and bone mineral density.
* Fibroscan: To determine the stiffness of the liver (liver elastography).
* Eye-examination: Visus, OPTOS, OCT og OCTA.
* Continuous blood glucose monitoring (CGM) Evaluation of glucose variability for at least 14 days. Most children and adolescent at our outpatient clinics use these as part of their regular regulation and treatment. If the participant normally uses a CGM-device, data on blood glucose variation from the past 90 days will be collected. If not a CGM-monitor will be placed on the upper arm and the participants will be instructed to wear it for the next 14 days.
* AX3: Physical activity for 7 days will be measured. Questionnaire Physical activity, Life quality
* Extended lungfunction

Medical history/journals Diabetes duration, treatment modality, insulin dosage, previous medication, episodes of diabetic ketoacidosis and hypoglycemia.

All earlier blood samples on: Hba1c, HDL, LDL, cholesterol. All earlier blood pressure, heart rate, weight, height, abdominal and hip circumference. Diabetic complication status: nephropathy, retinopathy, neuropathy or vascular complications. Data on current and prior asthma, atopy and eczema will be collected. Family history of type 2 diabetes, cardiovascular disease, asthma and atopy will be collected.

Insulin sensitivity Calculated using a validated score based upon Hba1c, waist circumference, fasting glucose and fasting insulin.

Participants will be recruited from the Paediatric Diabetes outpatient clinic at Steno Diabetes Center Copenhagen (SDCC) and Steno diabetes Center Sjælland (SDCS). All examinations and tests will be performed at SDCC. All children aged 6-18 years, with T1D for more than 12 months will be offered to participate. With a total of 950 T1D children/adolescent followed yearly at SDCC and 450 at SDCS the planned number of participants is realistic.

Sub-study I:

Insulin sensitivity (IS) has significant importance in T1D. The gold-standard measurement of IS is the hyperinsulinemic euglycemic clamp (HE clamp), a time-consuming procedure unfit for daily clinical practice. Thus, surrogate markers based on blood samples and anthropometric measurements have been developed. Only one of these surrogate markers is validated in youth with T1D and account for approximately 70 % of variance in IS. It has previously been demonstrated that lower IS, assessed by this surrogate marker, is associated with increased progression of arterial stiffness over time in youth with T1D. Arterial stiffness is associated with increased morbidity and mortality; thus, as IS is a modifiable risk factor it could serve as an instrument to reduce morbidity and mortality in T1D (17).

The hypothesis is that data from CGM devices can serve as a useful basis for constructing a surrogate marker for insulin sensitivity (IS), as CGM data provides comprehensive information on glucose metabolism and blood glucose patterns.

As a proof of concept, 14 pubertal boys (aged 14-18 years) will be invited to attend a second visit (Visit 1a), during which the gold-standard hyperinsulinemic-euglycemic (HE) clamp will be conducted. The clamp is performed in the morning after an overnight fast. A hyperinsulinemic state is induced through continuous insulin infusion for 2 hours and maintained until the end of the procedure.

Blood glucose is measured every 5-10 minute and glucose 20% is administrated based on these blood glucose measurements to keep a normal blood glucose level of 5-5.5 mmol/L. After approximately 2 hours, a steady state is achieved where the infusion of insulin and glucose balance one another. At this point glucose infusion rate (GIR) is measured and determines the glucose disposal rate (GDR). From the GDR the true physiological IS can be determined.

Data from CGM-devices and insulin administration 14 days prior to visit 1a will be analyzed in statistical models to predict IS, both direct measures (GDR) and assessed by the surrogate marker.

Statistics The methods applied to measure early markers of long-term diabetic complications both regarding arterial stiffness and the nerve system are all continuous parameters and no definitive cut offs between normal and early changes in children and adolescent are known. Therefore, sample size calculation for this study is not possible.

As described earlier, the SEARCH-study (7, 22) included some of the same outcome for evaluating cardiovascular-, nephrotic- and nerve system complications and showed statistically significant results with a number of 289 adolescents with T1D. The study plan to include 400 children and adolescent with T1D.

For descriptive data we will report frequency, mean (standard deviation) or median (interquartile range), as appropriate. Comparisons between relevant groups will be done for means with t-tests and medians with Mann-Whitney U-tests.

Linear regression models will be applied to assess the cross-sectional associations. Univariate and multivariable models will be used; adjustment will include risk factors and confounders based on prior evidence. In all analyses, model assumptions will be ascertained.

A two-sided p-value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* T1D>12 months
* 6-18 years old prior to inclusion
* Followed at the Pediatric Diabetes outpatient clinic at Steno Diabetes Center Copenhagen
* Speaks and reads Danish well enough to understanding the given oral and written information.
* There is a written consent from the guardianship holder/holders for the child.

Exclusion Criteria:

* T1D < 12 months
* Known cardiovascular disease
* Antihypertensive treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 400 children or adolescents with type 1 diabetes for more than 12 months. Age between 6-18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness in children and adolescent with type 1 diabetes (T1D) > 12 months and its association to glycemic control (current and past). | 15.01.2022-15.02.2024
  PWV is a measure of arterial stiffness (m/s) which can be done non invasively at bedside using a device called SphygmoCor CVMS machine (Atcor Medical, Sydney, Australia).
Peripheral neuropathy assed by DPN-check in children and adolescent with type 1 diabetes (T1D) > 12 months | 15.01.2022-15.02.2024
  Neuropathy assesed by DPN-check: Sural Nerve conduction velocity(m/s) of the Sural nerves by DPN-check.
Autonom neuropathy assed by Sudoscan in children and adolescent with type 1 diabetes (T1D) > 12 months | 15.01.2022-15.02.2024
  Neuropathy assesed by Sudoscan:
  Peripheral small-fiber sympathetic function (Sudoscan), measuring sudomotor function by electrochemical skin conductance (µS) in feet
Prevalence of cardivascular autonomic neuropathy assed by VagusDevice in children and adolescent with type 1 diabetes (T1D) > 12 months | 15.01.2022-15.02.2024
  The examination consists of 4 measures, all aimed at measuring heart rate. Measurements are taken for 5 minutes rest, change of position from lying to standing position, during deep breathing and by Valsalva (by breathing in a mouthpiece with a 40 mmHg resistance).

SECONDARY OUTCOMES:
The association between early markers of diabetic complications and glycemic control | 15.01.2022-15.02.2024
  Hba1c (mmol/mol)
The association between early markers of diabetic complications and glycemic control | 15.01.2022-15.02.2024
  Continous glucose monitoring (time in range (70-180mg/dL))

CONTACTS AND LOCATIONS:
Overall Officials: jesper johannesen, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No